CLINICAL TRIAL: NCT01406977
Title: An Open-label, Intra-patient Dose-escalation Study to Evaluate the Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of Multiple Infusions of BPS804 in Adults With Hypophosphatasia (HPP).
Brief Title: Dose Escalation Study to Evaluate the Safety and Tolerability of Multiple Infusions of BPS804 in Adults With Hypophosphatasia (HPP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Mereo BioPharma (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBPS804A2202; 2010-024013-31 (EudraCT Number)
Record Dates: First submitted 2011-07-29; First posted 2011-08-01 (Estimated); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Hypophosphatasia
Keywords: Hypophosphatasia; HPP; Rathbun's disease
MeSH Terms: conditions — Hypophosphatasia | interventions — setrusumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BPS804 dose escalation (Experimental): BPS804 IV Setrusumab given in escalating doses from 5mg/Kg to 20mg/Kg
  Interventions: Drug: BPS804

INTERVENTIONS:
Drug: BPS804

SUMMARY:
The purpose of the study is to determine tolerability, PK/PD and preliminary efficacy of BPS804 in adult patients with HPP treated with multiple escalating doses of BPS804.

This study will allow a comparison of several doses of the study drug within the first two weeks after administration and after a longer assessment period for the highest dose level to enable selection of dose ranges to be tested in subsequent studies in the HPP indication.

DETAILED DESCRIPTION:
This study was conducted and previously posted by Novartis. The record was transferred to Ultragenyx in February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 to 60 years of age in good health (other than pre-established clinical diagnosis of HPP) as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Previously established clinical diagnosis of HPP with confirmed ALPL mutation by genetic test and as manifested by:
* Serum alkaline phosphatase levels below the age-adjusted normal range and
* Radiologic evidence of osteopenia or osteomalacia or
* History of plasma PLP at least twice the upper limit of normal range or
* History of rickets, or history of premature loss of deciduous teeth, or bone deformity consistent with osteomalacia or past rickets, or past non-traumatic fracture, pseudofracture, or non-healing fracture.
* 25-(OH) vitamin D3 serum level of ≥20 ng/mL.
* Normocalcemia with serum calcium ≥8.5 mg/dL and ≤10.2 mg/dL and normal phosphate levels (2.4 - 4.1 mg/dL) (or according to local laboratory ranges).

Exclusion Criteria:

* A history of clinically significant ECG abnormalities.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin and for skeletal malignancies see below), within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* History of skeletal malignancies or bone metastases at any time.
* History of external beam radiation to the skeleton.
* Open epiphyses as judged by the Investigator based on previous clinical assessments.
* Patients with suspected neural foraminal stenosis (e.g., at cervical, spinal, or lumbar site) as judged by the Investigator which could be caused by disc herniation and are described as sciatic pain, tingling, burning sensation with numbness and/or weakness.
* History of or concomitant diseases such as hypo-/hyperparathyroidism, hypo-/hyperthyroidism, Pagets disease, previous neck surgery involving partial or complete thyroidectomy and abnormal thyroid function or thyroid disease or other endocrine disorders or conditions.
* Treatment with any anti-resorptive medication (e.g., oral and/or injectable), bisphosphonates and/or teriparatide (e.g., ForteoTM) within the last 6 months.
* Exposure to blood products or monoclonal antibodies within previous 12 months.
* Any deformation of the spine (e.g., severe scoliosis, ankylosing spondylitis) or the hip which would preclude proper acquisition of lumbar spine or hip BMD by DXA.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
The number (percent) of patients experiencing adverse events or serious adverse events | 141 days following initial investigational product administration
Change from baseline in primary serological bone biomarkers | 141 days following initial investigational product administration

SECONDARY OUTCOMES:
Characterization of the pharmacokinetic profile of BPS804: area under the plasma concentration-time curve (AUC) | 1, 29 and 141 days following initial investigational product administration
Characterization of the pharmacokinetic profile of BPS804: observed maximum plasma concentration following drug administration (Cmax) | 1, 15 and 29 days following initial investigational product administration
Characterization of the pharmacokinetic profile of BPS804: time to reach the maximum concentration (Tmax) | 1, 15 and 29 days following initial investigational product administration
Change from baseline in secondary biomarkers | 141 days following initial investigational product administration
The number (percent) of patients developing anti-BPS804 antibodies | 141 days following initial investigational product administration

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (1):
- Mereo BioPharma 3 Ltd Investigative Site, Würzburg, Germany

REFERENCES:
- [Derived] Seefried L, Baumann J, Hemsley S, Hofmann C, Kunstmann E, Kiese B, Huang Y, Chivers S, Valentin MA, Borah B, Roubenoff R, Junker U, Jakob F. Efficacy of anti-sclerostin monoclonal antibody BPS804 in adult patients with hypophosphatasia. J Clin Invest. 2017 Jun 1;127(6):2148-2158. doi: 10.1172/JCI83731. Epub 2017 Apr 24. PMID 28436937